CLINICAL TRIAL: NCT07271628
Title: Evaluation of the Moisturizing Effect of Study Product AV0018B and the Persistence of This Effect After Repeated Applications, Compared to an Untreated Control Area.
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: MINIREGETA
Record Dates: First submitted 2025-11-25; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Dry Skin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AV0018B application
  Interventions: Other: Cosmetic product AV0018B
- No AV0018B application

INTERVENTIONS:
Other: Cosmetic product AV0018B — Cosmetic spray product AV0018B. The product is sprayed 6 times per day for 7 days. The spraying of about 3 sec is done on the inner and posterointernal side of the concerned forearm (according to randomization)
  Groups: AV0018B application

SUMMARY:
This study is a monocentric, intra-individual, controlateral design study, on the internal and posterointernal side of the forearms, to evaluate the moisturizing effect of study product AV0018B and of the persistence of this effect after repeated applications for 7 days, compared to a control area with no application of study product.

The study takes place over a 8-day period and involves 2 visits :

* Inclusion visit: Day 1 (1timepoint (Time 1) before any study product application)
* End-of-study visit: Day 8 (2 timepoints : Time 2 : 12±2h after last application , and Time 3 : 8±4h after Time 2)

ELIGIBILITY:
Inclusion Criteria:

* Females
* Aged 20 to 55 years, inclusive
* Phototype I to V, inclusive
* Low hairiness and absence of prominent veins on the internal and posterointernal side of the forearms.
* No shaving/hair removal of forearms
* Dehydrated forearms, with HI ≤ 35 (posterointernal side of the forearms)
* Not taking part in another clinical research study.
* Having signed the consent form.
* Having health insurance.

Exclusion Criteria:

Population:

* Pregnant, breastfeeding women.
* Subjects declaring to have hot flushes.
* With sunburn on forearms.
* Frequently washing their forearms for professional reasons or out of habit.
* Application of keratolytic and/or self-tanning products to the upper limbs in the 4 weeks prior to inclusion.
* Application of skin care (Hydrating, nourishing) or exfoliating products to the upper limbs in the 2 weeks prior to inclusion.
* Application of water or hygiene products to the upper limbs since the last wash on the evening before inclusion.
* Participating in another study on the forearms (not including kinetics studies) in the 2 weeks prior to inclusion.
* Participating in a kinetics study on the forearms in the 48 hours prior to inclusion.
* Subjects unable to comply with the protocol requirements.
* Subjects deprived of freedom through a legal or administrative decision, or in care or under legal guardianship.

Diseases:

* History of allergy to any of the investigational product ingredients
* Skin lesions or skin disease on the hands, arms and forearms.
* Type 1 diabetes.
* Unresolved viral hepatitis.
* Chronic cardiovascular, endocrine, rheumatological and urogenital system and non-stabilized neuropsychiatric disorders (treatment started less than 2 months ago).
* Acute pathology (infectious, inflammatory).
* Dermatological condition or skin lesion on the top of the cheekbone liable to interfere with the samplings according to the investigator's opinion.
* Any skin characteristic on the top of the cheekbone incompatible with the samplings (raised nevus, etc.) according to the investigator's opinion.

Treatments:

* Ongoing local treatment (dermocorticosteroids, retinoids, antibiotics, antifungals, etc.) or treatment applied in the 7 days prior to inclusion.
* Ongoing oral antibiotic and/or anti-inflammatory (steroid and non-steroid) or treatment taken for more than 5 consecutive days in the week before inclusion.
* Oral treatment (cardiovascular, endocrine, rheumatological, urogenital, neuropsychiatric, immunosuppressant) started in the 2 months prior to inclusion.
* Any local treatment applied to the face in the week preceding the inclusion visit
* Application of water, any rinsed or leave-on cleansing or care product on the face after the last wash performed the day before the inclusion visit

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects will be recruited from the panel of the centre (corresponding to an internal computer database whose software has been declared to the Commission Nationale Informatique et Libertés (CNIL)).
  If necessary, a local announcement/advertising will be done. The subjects corresponding to eligibility criteria may receive a phone call, a letter or an e-mail proposing to participate to the clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Cutaneous Capacitance | - Visit 1 : Day 1 - Time 1 - Visit 2 : Day 8 - Time 2 (12±2hours after last application) and Time 3 (8±4hours after Time 2)
  Cutaneous capacitance is measured by Corneometry at posterointernal sides of forearms.

SECONDARY OUTCOMES:
Illustrative Photographs | - Visit 1 : Day 1 - Time 1 - Visit 2 : Day 8 - Time 2 (12±2hours after last application) and Time 3 (8±4hours after Time 2)
  Photographs on posterointernal sides of forearms using the calibrated video camera and Moisture Map® tool, for illustrative purpose only.

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Research Center, Toulouse, France, France